CLINICAL TRIAL: NCT01070758
Title: Treatment With Lanreotide Autogel (Somatostatin Analogue) in Patients With Congenital Hyperinsulinism of Infancy Already Treated With Somatostatin Analog by Pump
Brief Title: Lanreotide Autogel Treatment of Patients With Congenital Hyperinsulinism of Infancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Dalit Modan, Pediatric Endocrinologist, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-10-7165-DM-CTIL
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Congenital Hyperinsulinism
Keywords: Congenital hyperinsulinism; Somatostatin analog; Lanreotide autogel; Hypoglycemia
MeSH Terms: conditions — Congenital Hyperinsulinism; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Single arm open label study
  Interventions: Drug: Lanreotide autogel

INTERVENTIONS:
Drug: Lanreotide autogel — The dose of Lan-ATG will be calculated according to the surface area of the patient. The dose used in adults is usually 60 mg injection once a month, and we will adapt the patient's dose according to the body surface area and also according to the daily dose of Octreotide used with the pump. The starting dose will be 40 mg/m².
  Other Names: Somatuline autogel

SUMMARY:
The purpose of our study is to evaluate the efficacy and safety of Lanreotide Autogel in children with congenital hyperinsulinism already treated with Octreotide by pump.

Congenital hyperinsulinism is a genetic disorder characterized by inappropriate insulin secretion resulting in persistent hypoglycemia (low blood sugars. Patients exposed to recurrent hypoglycemic episodes are at increased risk of developmental disorders, so identification and prompt management of patients are essential. Many patients are treated with the somatostatin analog Octreotide which is administered by continuous infusion using a pump (we use an insulin pump). This treatment may pose a huge burden and be stressful for patients and families as it demands intensive daily care. In an effort to simplify the daily care of our patients and improve their quality of life we will study the efficacy and safety of Lanreotide Autogel - a long-acting somatostatin analog that can be administered by injection once a month

DETAILED DESCRIPTION:
The purpose of our study is to evaluate the efficacy and safety of Lanreotide Autogel in children with CHI already treated with Octreotide by pump.

Patients and methods. Congenital hyperinsulinism (CH) is a genetic disorder characterized by dysregulated insulin secretion resulting in persistent hypoglycemia. Identification and prompt management of patients are essential, as patients exposed to recurrent hypoglycemic episodes are at increased risk of developmental disorders. Many patients are treated with the somatostatin analog Octreotide which is administered by continuous infusion using a pump. This treatment may pose a huge burden and be stressful for patients and families as it demands intensive daily care. In an effort to simplify the daily care of our patients and improve their quality of life we will study the efficacy and safety of Lanreotide Autogel(Lan-ATG)- a long-acting somatostatin analog that can be administered by injection once a month.

This trial will include children with CH, who are treated with Octreotide by pump. We believe that children older than 2 years old will benefit most from this therapy. At this age, some of the parents encounter technical problems with the pump, as the children are prone to play with the pump and take out the needles. It's also very difficult to place the children in day care, because they need continuous follow up.

The dose of Lan-ATG will be calculated according to the surface area of the patient. The dose used in adults is usually 60 mg and we will adapt the patient's dose according to the body surface area and also according to the daily dose of Octreotide used with the pump. The starting dose will be 40 mg/m².

The patients will be gradually weaned from the pump following the first injection of Lan-ATG (10% decrease every 3-4 days for a total of a month).

Every patient will serve as his/her own control.

The following examinations will be done in every child:

1. Continuous blood glucose monitoring during 72 hours with a glucosensor, to exclude asymptomatic hypoglycemia - once in 6 months.
2. Growth velocity every 3 months.
3. Bone age once a year.
4. Routine laboratory tests (biochemistry, CBC and thyroid function tests) every six months.
5. Biliary US once in 6 months. During the follow up we will try to expand the distance between injections, based on our knowledge that most of the patients with CH are known to enter remission after the age of 4-5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-8 years,
* Diagnosed with congenital hyperinsulinism,
* Treated by Octreotide continuous infusion (pump).

Exclusion Criteria:

* Family not interested in participating.

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2010-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Euglycemia as recorded by Continuous Glucose Monitoring System (CGMS) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dalit Modan, M.D., Principal Investigator — Sheba Medical Ceter, Tel-Hashomer, Israel
Locations (1):
- Pediatric Endocrinology Unit, Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Derived] Modan-Moses D, Koren I, Mazor-Aronovitch K, Pinhas-Hamiel O, Landau H. Treatment of congenital hyperinsulinism with lanreotide acetate (Somatuline Autogel). J Clin Endocrinol Metab. 2011 Aug;96(8):2312-7. doi: 10.1210/jc.2011-0605. Epub 2011 Jun 22. PMID 21697252